CLINICAL TRIAL: NCT03331510
Title: Change of Strength and Range of Motion in Arthroscopic Latarjet Procedure - A Prospective Trial Involving the Four Muscles Altered
Brief Title: Prospective Strength Measurement Involving Muscles Altered In Arthroscopic Latarjet
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Etzel Clinic (Other)
Responsible Party: Principal Investigator, Daniel Smolen, MD, MD, Etzel Clinic
Other Study IDs: Prospective Strength Latarjet
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Shoulder Instability
Keywords: Shoulder, Instability, Latarjet, Dislocation, Strength
MeSH Terms: conditions — Joint Dislocations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Strength testing before and after arthroscopic Latarjet — After patients, based on the ISI-Score, were assigned to treat their shoulder instability with an arthroscopic Latarjet procedure, they are eligible for this study. Strength of different involved muscles, as well as ROM will be measured before and at several time points after surgery.

SUMMARY:
Open and arthroscopic Latarjet procedures are used to treat shoulder instability as primary and salvage procedures. During surgery the coracoid process is detached and repositioned to the anterior glenoid through a subscapularis split and fixed in place, resulting in an enlarged glenoid and therefor articular surface. However, before this is done, the pectorals minor, which inserts at the coracoid process, has to be detached and is left without further treatment. Moreover, the conjoint tendon, the origin of the short head of the biceps and coracobrachialis, is repositioned with the coracoid and therefor distalized and medialized.

No study currently followed up on the strength of the muscles altered. The aim of this study is therefor, to prospectively measure range of motion and strength of the operated shoulder at different time points pre- and postoperatively, comparing it with the healthy shoulder in each individual.

DETAILED DESCRIPTION:
Strength, range of motion and stability will be assessed pre-operatively and at 6 weeks, 12 weeks, 6 months, 12 months and 24 months post-operatively. Next to standard radiological follow up, including X-ray, arthrographic computed tomography as well as arthrographic magnetic resonance imaging, specific shoulder scores will be utilised. Strength for general shoulder motion as well as specifically for the subscapularis, the pectorals minor, the coracobrachialis and the biceps will be measured with a shoulder dynamometer. Data will be analysed and published.

ELIGIBILITY:
Inclusion Criteria:

* Patients who experienced at least one shoulder dislocation.
* Patients who are willing to participate in the study
* Patients who receive arthroscopic Latarjet procedure for treatment of glen-humeral instability
* Patients who are at least 18 years old.
* Patients with an ISI-Score of at least 4 points.

Exclusion Criteria:

* Patients older than 50 or younger than 18 years of age.
* Patients with painful unstable (multidirectional) instability
* Patients with congenital defects of the bones involved (humerus, scapula).
* Patients with an ISIS of smaller 4 points.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Patients with shoulder instability or shoulder dislocations, treated with arthroscopic Latarjet at the Etzelclinic will be enrolled in consideration of the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Strength | 24 months
  Strength for different muscles involved in shoulder movement is measured pre- and post-operatively for the operated shoulder and the contralateral side. Strength will be measured in Kilogramm with a shoulder dynamometer. Scale range is assumed to be between 0 and 25 kg, higher values postoperatively indicate better outcome. Measurements will be undertaken for the subscapularis in internal rotation at 0 and 90 degrees; for the muscles attached to the conjoint tendon (short head of the biceps and coracobrachialis) in 45 degree shoulder flexion, while resistance will be applied on the flexing forearm. The pectoralis minor measurment will be undertaken through applying pressure against the protracting shoulder. Furthermore, standard strength measurements will be undertaken in 90 degree shoulder flexion and abduction, applying resistance against the hand, and in 0 degree internal as well as external rotation with a flexed elbow.

SECONDARY OUTCOMES:
Range of Motion | 24 months
  Range of Motion of the operated shoulder and the contralateral side is measured pre-and post-operatively. Outcome measure will be in degree of range of motion, with higher numbers indicating greater range of motion.
Stability | 24 months
  Stability of the operated shoulder is evaluated objectively and subjectively utilising different specific scores.

IPD SHARING:
Plan to Share IPD: Yes
To discuss and evaluate results as well as drafting the manuscript, IPD might be shared with other researchers.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: As soon as data of each patient involved is collected, it will possibly be shared with participating researchers and experienced advisors, until final manuscript is drafted.
Access Criteria: Personal (eye to eye)